CLINICAL TRIAL: NCT03509441
Title: Early MRI Detection of Myocardial Deterioration as a Preventive, Disease Staging, and Prognostic Biomarker in Insulin Resistance
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Rajesh Dash, MD PHD, Asst Prof-Med Ctr Line, Stanford University
Other Study IDs: 31279
Record Dates: First submitted 2017-05-08; First posted 2018-04-26 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cardiomyopathies; Insulin Resistance; Non-ischemic Cardiomyopathy; Cardiac Fibrosis; Diabetes
Keywords: South Asian; Insulin Resistance; Cardiac Fibrosis; MRI; Diabetes; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators will probe individual patient risk based on initial cardiac fibrosis measurements. In insulin resistance, the degree of fibrosis may be out of proportion to disease severity, pointing to a genetic predisposition for increased cardiac cell dropout (i.e. apoptosis) and replacement fibrosis. To address this idea, the investigators will collect and store peripheral blood samples from every patient, identify those with high and low fibrosis levels, and then select patients with disproportionately high fibrosis levels given their disease burden. Induced pluripotent stem cell-derived cardiomyocytes (iPSC- CMs) will then be generated. The iPSC-CMs will be tested, in vitro, for drug sensitivity, susceptibility to apoptotic stimuli, and the propensity to produce pro-fibrotic cytokine activation. In this manner, the investigators will study the individual patient's myocardial cell features that increase the risk of cardiac fibrosis and the subsequent adverse outcomes that ensue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- South Asians with Insulin Resistance: 125 patients (anticipated)
- South Asians without Insulin Resistance: 125 patients (anticipated)

SUMMARY:
The purpose of this study is to evaluate the relationship between insulin resistance (IR) and myocardial tissue abnormalities. The study will focus on a patient population, South Asians, with a high prevalence of IR.

DETAILED DESCRIPTION:
Cardiac fibrosis has been linked to adverse outcomes in non-ischemic cardiomyopathy. Fibrosis is also detectable in diabetic patients, but does not appear to closely track with insulin sensitivity. Hence, fibrosis may be an independent risk factor for adverse outcomes in IR and diabetic patients. As a result, a critical need exists to develop a non-invasive tool to identify and treat the highest-risk patients. Early detection of cardiac fibrosis and other CMR- detectable abnormalities in IR patients may help to 'stage' a patient's disease process and future risk of events, ultimately leading to an adjustment in the aggressiveness of their medical management and long-term monitoring accordingly. This project is aimed at reducing the mortality and morbidity associated with insulin resistance and diabetes, and the investigators believe this project could have a transformative impact on long-term diabetic care and shed new light upon the biology of diffuse cardiac fibrosis in insulin resistance and diabetes and its role in shaping the long-term cardiovascular risk for these patients.

ELIGIBILITY:
Inclusion Criteria:

- South Asian

Exclusion Criteria:

* Pregnant women
* Patients with prior diagnoses of diabetes
* Patients on insulin therapy
* Patients with known coronary heart disease or other non-ischemic cardiomyopathies

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: South Asians between the age of 20 and 60 who have no active coronary heart disease or other non-ischemic cardiomyopathies
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Identifying patients with high fibrosis levels using peripheral blood samples | Blood samples drawn once at baseline visit
  The investigators will collect and store peripheral blood samples from every patient, identify those with high and low fibrosis levels using our described protocol, and then select patients with disproportionately high fibrosis levels given their disease burden.
  The investigators can test for the level of fibrosis by generating induced pluripotent stem cell-derived cardiomyocytes (iPSC- CMs) from these collected blood samples. These iPSC-CMs will be tested, in vitro, for drug sensitivity, susceptibility to apoptotic stimuli, and the propensity to produce pro-fibrotic cytokine activation- all factors which will help the investigators determine fibrosis levels.
Insulin Sensitivity measured by OGTT | OGTT done at baseline/ first visit
  An oral glucose tolerance test with insulin measurement (OGTT) will be performed for all the patients. The investigators will draw blood to determine a fasting glucose measurement, and then the patients will be given a 75 g glucose solution to drink. Blood samples will be collected at serial time points (30 minutes, 60 minutes, 120 minutes) after ingestion of this liquid to determine blood glucose and insulin levels. The OGTT will help investigators determine the patient's degree of insulin sensitivity.
Insulin Sensitivity measured by Fasting Lipid Panel | Lipid Panel done at baseline/ first visit
  Baseline fasting lipids will be assessed to calculate a TG/HDL-C ratio, which also correlates with the degree of insulin sensitivity or lack thereof. These results will be correlated to the insulin sensitivity assessment performed by the OGTT.
Left ventricular volume | CMR done at baseline visit
  Cardiac MRI/ CMR done to noninvasively image heart and determine volume of left ventricle
Left ventricular mass | CMR done at baseline visit
  Cardiac MRI/ CMR done to noninvasively image heart and determine mass of left ventricle
Ejection fraction % | CMR done at baseline visit
  Cardiac MRI/ CMR done to noninvasively image heart and determine ejection fraction
Myocardial tagging for strain analysis | CMR done at baseline visit
  Cardiac MRI/ CMR done to noninvasively image heart and assess ventricular function through myocardial tagging. By modulating the magnetization gradient of the MRI prior to acquiring images, any parts of the heart which are not contracting can be identified. These images will be analyzed via strain analysis for such abnormalities in function
Assessing diffuse fibrosis via T1 mapping | CMR done at baseline visit
  A CMR technique called T1 mapping will be performed to calculate level of extracellular volume (ECV), which helps with the quantification of diffuse fibrosis
Assessing level of edema via T2 mapping | CMR done at baseline visit
  A CMR technique called T1 mapping will be performed assess amount of edema in the heart

SECONDARY OUTCOMES:
Collagen turnover assessment | Blood drawn at baseline visit
  Patients will have blood drawn for serum measurement of propeptides of several procollagens to determine the level of collagen turnover
Endothelial Function | 15 minute procedure done at baseline visit
  The investigators will also measure endothelial function using the endoPAT device, which employs noninvasive measurement of finger arterial pulsatile volume changes as a measure of endothelial function. This test takes approximately 15 minutes and is noninvasive.
Urine test for albumin levels | One urine test done at baseline visit
  24 Hour urine test for assessment of albumin levels
Urine test for creatinine levels | One urine test done at baseline visit
  24 Hour urine test for assessment of creatinine levels

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Dash, MD, PhD, Principal Investigator — Stanford University; Abha Khandelwal, MD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No